CLINICAL TRIAL: NCT03909139
Title: Prospective PROMs Outcomes in Arthroscopic Acetabular Labral Repair With and Without Application of Platelet-Rich Plasma (PRP) Harvested From the Body of the Ilium
Brief Title: Use of BMAC With Hip Arthroscopy Treatment of FAI and Labral Tear
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Scott D Martin, Principal Investigator, Director, Joint Preservation Service, Director, MGH Sports Medicine Fellowship, Massachusetts General Hospital
Other Study IDs: 2019P002191
Record Dates: First submitted 2018-06-11; First posted 2019-04-09 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Acetabular Labrum Tear; Femoro Acetabular Impingement; Chondral Defect; Bone Marrow Aspirate Concentrate; Mesenchymal Stromal Cell
Keywords: Acetabular Labrum Tear; Femoro Acetabular Impingement; Chondral Defect; Bone Marrow Aspirate Concentrate; Mesenchymal Stromal Cell; Chondrolabral Junction; Osteoarthritis; Femoroacetabuloplasty; Hip Arthroscopy; BMAC
MeSH Terms: conditions — Femoracetabular Impingement; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Bone marrow is aspirated then centrifuged. From the centrifuged sample, the buffy coat layer (layer of cells, found between the red blood cells and the plasma layers) is removed. The buffy coat layer contains mesenchymal stromal cells. This sample of centrifuged, concentrated mesenchymal stromal cells is called BMAC or Bone Marrow Aspirate Concentrate. The BMAC will be injected into the intra-articular space.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- BMAC Application: Patients age 18 or older with evidence consistent with a tear of the acetabular labrum and breakdown of the chondrolabral junction and consent to arthroscopic labral tear repair.
  BMAC application at the time of arthroscopic labral repair.
  Interventions: Biological: BMAC
- No BMAC Application: Patients age 18 or older with evidence consistent with a tear of the acetabular labrum and breakdown of the chondrolabral junction and consent to arthroscopic labral tear repair.
  No BMAC application at the time of arthroscopic labral repair.

INTERVENTIONS:
Biological: BMAC — A bone marrow biopsy needle will be inserted through an arthroscopy portal and directed to the acetabuloplasty site. Bone marrow is aspirated then centrifuged. From the centrifuged sample, the buffy coat layer (layer of cells, found between the red blood cells and the plasma layers) is removed. The buffy coat layer contains mesenchymal stromal cells. This is called BMAC or Bone Marrow Aspirate Concentrate. The BMAC will be injected into the intra-articular space.
  Groups: BMAC Application

SUMMARY:
Femoro-acetabular impingement is a well known cause of damage to the acetabular labrum and chondrolabral junction. Additionally, it has been proposed that disruption of hip biomechanics resulting from a labral tear causes a faster progression towards osteoarthritis (OA). This progression has been observed to begin with breakdown of the chondrolabral junction with later development of diffuse osteoarthritis. Use of hip arthroscopy has increased dramatically in recent years to treat symptomatic labral tears and potentially avoid the morbidity and cost associated with hip osteoarthritis.

Correction of labral pathology presents a technical challenge and many techniques currently exist. Increased understanding of the structure-functional relationship dictated by labral anatomy has led to the development of methods aimed at restoring functional anatomy by re-establishing the labrum's native position and contour on the rim of the acetabulum. Therefore, akin to repairing a torn meniscus in the knee, restoring the anatomic footprint of a torn labrum will reconstitute normal joint biomechanics.

Despite the advances in techniques for labral repair, strategies for mitigating or repairing damage to the chondrolabral junction do not yet exist. This area has been shown to consist of hyaline and fibro cartilage. Many techniques for cartilage repair exist, although most are not feasible due to technical challenges specific to the hip joint.

The management of articular cartilage defects is one of the most challenging clinical problems for orthopaedic surgeons. Articular cartilage has a limited intrinsic healing capacity, and pathology frequently results in gradual tissue deterioration. Currently, the standard surgical intervention for end-stage degenerative joint pathology is total joint replacement. Early surgical interventions for symptomatic cartilage lesions including cell based therapies such as autologous chondrocyte implantation (ACI), bone marrow aspirate concentrate (BMAC) implantation, or microfracture have been suggested to restore normal joint congruity and minimize further joint deterioration. Techniques such as ACI, which have been successfully used in the knee joint, have limited application in the hip due to the technical difficulties of open procedures.

DETAILED DESCRIPTION:
The acetabular labrum is a wedge shaped fibrocartilage structure attached to the acetabular rim. It is continuous with the transverse acetabular ligament at the inferior aspect of the acetabulum. The medial aspect of the labrum abuts the acetabulum to form the chondrolabral junction.

Anatomic labral refixation aims to preserve healthy tissue and restore native joint anatomy and biomechanics. Labral tears that are caused by Femoro-Acetubular Impingement (FAI) require concomitant correction of bony cam lesions, pincer lesions, or both to prevent reinjury of the labrum. However, repair has not yet been proven to mitigate the osteoarthritic accelerating effects of labral tears. Many patients presenting with hip pain in the third and fourth decade of life already have osteoarthritic changes seen at the time of arthroscopy. Restoring the biomechanics of the joint via labral repair does not reverse this damage and investigating methods to repair early osteoarthritis is important to the future of hip arthroscopy.

Bone marrow aspirate concentrate (BMAC) has been used effectively in many joints for the management of chondral defect repair. As an alternative to the aforementioned chondral treatment modalities, BMAC treatment does not require multiple procedures or additional waiting time for treatment completion.

Within the technical constraints of the hip joint, bone marrow aspirate concentrate is feasible and potentially efficacious option for the treatment of chondral defects. Late stage hip osteoarthritis is a known factor implicated in poor outcomes in both the surgical and non-surgical treatment options available for chondral defect management. Preventing late stage hip osteoarthritis is paramount to decrease these poor outcomes and improve the patient's quality of life. Early and effective intervention with modalities that afford patients little to no drawbacks, like BMAC treatment, are necessary to achieve these goals.

This is a prospective study which will enroll 400 adult subjects with evidence of an acetabular labrum tear and pincer or cam deformity. Labral tears will be diagnosed by clinical exam and positive magnetic resonance arthrogram (MRA) findings. Pincer deformity is diagnosed with standard antero-posterior radiographs of the pelvis, and cam deformity is diagnosed with antero-posterior and lateral radiographs.

Administration of diagnostic modalities is independent of study protocol as they are routine standard of care. Upon diagnosis, eligible potential subjects will be approached for study enrollment. After consent, enrolled subjects will undergo arthroscopic labral repair using a capsular chondrolabral preservation technique with or without BMAC based on intra-operative findings. The decision to use BMAC is made intra-operatively; therefore the patients are consented for the BMAC prior to surgery. If the chondrolabral junction shows advanced arthritis or the absolute absence of wear the BMAC is unnecessary and not used. This surgery in the absence of BMAC is considered routine practice and standard of care. Subjects will follow-up at routine post-operative intervals of 3 months, 6 months, 12 months, and annually thereafter to monitor progress.

Interval Results:

Martin SD, Kucharik MP, Abraham PF, Nazal MR, Meek WM, Varady NH. Functional Outcomes of Arthroscopic Acetabular Labral Repair with and without Bone Marrow Aspirate Concentrate [published online ahead of print, 2021 Oct 14]. J Bone Joint Surg Am. 2021;10.2106/JBJS.20.01740. doi:10.2106/JBJS.20.01740

ELIGIBILITY:
Inclusion Criteria and Rationale:

1. Age 18 or older: patients of any age have the capacity to potentially benefit from labral repair
2. Symptoms consistent with a tear of the acetabular labrum (i.e., catching, clicking, popping, pain with sitting, episodic pain, pain with hip flexion, adduction, and/or internal rotation): asymptomatic labral tears do exist in the general population however there is not definitive evidence to suggest treatment of asymptomatic tears is beneficial.
3. Symptoms not due to some other acute process in or around the hip (including septic arthritis, osteonecrosis, hemarthrosis, iliotibial band syndrome, fractures of the femoral neck or head, fractures of the acetabulum, greater trochanteric pain syndrome, sacroiliac joint pain, piriformis syndrome, low back pain associated with hip pain and not knee nor acute low back injury): certain conditions are not treatable by either arthroscopy or physical therapy. Some of these conditions can be managed with physical therapy but not arthroscopy.
4. Availability of hip radiographs and magnetic resonance imaging (MRI and/or MRA): needed to assess eligibility
5. Evidence of labral tear on MRI and/or MRA: documentation of acetabular labrum tear
6. Willingness to participate and ability to understand and sign informed consent document: ability to understand study and consent willingly
7. Returning subjects enrolled in protocol 2017P001391/PHS

Exclusion Criteria and Rationale:

1. Non-English speaking subjects: PROMs are only validated in English.
2. Systemic infection: surgery is generally contraindicated when systemic infection is present.
3. Systemic heparinization: the vascularity of the bone and adjacent tissues is significant, posing a potential problem for bleeding when the patient is anti-coagulated.
4. Pregnant women/fetuses: although surgery can be performed on pregnant women, pregnant women are excluded under federal regulations.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This is a prospective study which will enroll adult subjects with evidence of an acetabular labrum tear. These subjects will be enrolled consecutively using the aforementioned criteria until we hit our enrollment of 300 subjects.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-09-06 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change iHOT--33 Surveys from preoperative to various postoperative timepoints | Baseline (pre-operative), 3 months, 6 months, 12 months, and annually thereafter
  Full Name of Outcome: International Hip Outcome Tool--33 Questions
  Purpose: Validated Hip Patient Reported Outcome Measurements (PROMs) to assess the patient's functional outcomes post-surgery.
  Scale of iHOT-33:
  Min: 0 Max: 100
  No standardized scoring categories (i.e. excellent, good, fair, poor).
  Higher score indicates better hip functionally.
  No subscores or subscales

SECONDARY OUTCOMES:
Change HOS Surveys from preoperative to various postoperative timepoints | Baseline (pre-operative), 3 months, 6 months, 12 months, and annually thereafter
  Full Name of Outcome: HOS--Hip Outcome Score, which consists of two subscores: Hip Outcome Score-Activity of Daily Living (HOS-ADL), Hip Outcome Score-Sports Sub-scale (HOS-SSS)
  Purpose: Validated Hip Patient Reported Outcome Measurements (PROMs) to assess the patient's functional outcomes post-surgery.
  Scale of HOS--ADL:
  Min: 0 Max: 68
  Converted to a percentage, by dividing patient's score by 68.
  No standardized scoring categories (i.e. excellent, good, fair, poor).
  Higher score indicates better hip functionally.
  Scale of HOS--SSS:
  Min: 0 Max: 36
  Converted to a percentage, by dividing patient's score by 36.
  No standardized scoring categories (i.e. excellent, good, fair, poor).
  Higher score indicates better hip functionally.
Change NAHS Surveys from preoperative to various postoperative timepoints | Baseline (pre-operative), 3 months, 6 months, 12 months, and annually thereafter
  Full Name of Outcome: Non-Arthritic Hip Score (NAHS)
  Purpose: Validated Hip Patient Reported Outcome Measurements (PROMs) to assess the patient's functional outcomes post-surgery:
  Scale of NAHS:
  Min: 0 Max: 100
  No standardized scoring categories (i.e. excellent, good, fair, poor).
  Higher score indicates better hip functionally.
  No subscores or subscales.
Change LEFS Surveys from preoperative to various postoperative timepoints | Baseline (pre-operative), 3 months, 6 months, 12 months, and annually thereafter
  Full Name of Outcome: Lower Extremity Functional Scale (LEFS)
  Purpose: Validated Hip Patient Reported Outcome Measurements (PROMs) to assess the patient's functional outcomes post-surgery.
  Scale of LEFS:
  Min: 0 Max: 80
  Converted to a percentage, by dividing patient's score by 80.
  No standardized scoring categories (i.e. excellent, good, fair, poor).
  Higher score indicates better hip functionally.
  No subscores or subscales
Change mHHS Surveys from preoperative to various postoperative timepoints | Baseline (pre-operative), 3 months, 6 months, 12 months, and annually thereafter
  Full Name of Outcome: modified Harris Hip Score (mHHS)
  Purpose: Validated Hip Patient Reported Outcome Measurements (PROMs) to assess the patient's functional outcomes post-surgery.
  Scale of mHHS:
  Min: 0 Max: 100
  Scoring of mHHS:
  Excellent: 90--100 Good: 80--89 Fair: 70--79 Poor: <70
  Higher score indicates better hip functionally.
  No subscores or subscales.
Change RAND-36 Surveys from preoperative to various postoperative timepoints | Baseline (pre-operative), 3 months, 6 months, 12 months, and annually thereafter
  RAND-36 Measure of Health-Related Quality of Life (RAND 36 or SF 36):
  The most widely used health-related quality-of-life survey instrument
  Consists of 36 questions that assess eight components of health: physical functioning, role limitation due to physical health problems, role limitations due to emotional problems, social functioning, emotional well-being, energy/fatigue, pain, and general health perceptions, with a simple mean of these responses ranging from 0 to 100, with 100 representing the best possible quality-of-life score.
Degree of Improvement on Hip VAS Pain Score | Baseline (pre-operative), 3 months, 6 months, 12 months, and annually thereafter
  At routine follow-up visits patients will be asked to rate hip pain using the VAS (Visual Analog Scale) Score
  Min: 0--no pain Max: 10--worst pain experienced in their life
  Increments of 1.
  Categories:
  1--3: mild pain 4--6: moderate pain 7--10: severe pain
Patient Satisfaction Questionnaires | 12 months and annually thereafter
  Three Yes/No Questions:
  1. Are you satisfied with the treatment you received?
  2. Are you satisfied with the treatment regimen that you were given?
  3. If given the choice in the future, would you choose the same treatment?

CONTACTS AND LOCATIONS:
Overall Officials: Scott D Martin, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH, Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cotten A, Boutry N, Demondion X, Paret C, Dewatre F, Liesse A, Chastanet P, Fontaine C. Acetabular labrum: MRI in asymptomatic volunteers. J Comput Assist Tomogr. 1998 Jan-Feb;22(1):1-7. doi: 10.1097/00004728-199801000-00001. PMID 9448753
- [Background] Register B, Pennock AT, Ho CP, Strickland CD, Lawand A, Philippon MJ. Prevalence of abnormal hip findings in asymptomatic participants: a prospective, blinded study. Am J Sports Med. 2012 Dec;40(12):2720-4. doi: 10.1177/0363546512462124. Epub 2012 Oct 25. PMID 23104610
- [Background] Ganz R, Parvizi J, Beck M, Leunig M, Notzli H, Siebenrock KA. Femoroacetabular impingement: a cause for osteoarthritis of the hip. Clin Orthop Relat Res. 2003 Dec;(417):112-20. doi: 10.1097/01.blo.0000096804.78689.c2. PMID 14646708
- [Background] Field RE, Rajakulendran K. The labro-acetabular complex. J Bone Joint Surg Am. 2011 May;93 Suppl 2:22-7. doi: 10.2106/JBJS.J.01710. PMID 21543684
- [Background] Song Y, Ito H, Kourtis L, Safran MR, Carter DR, Giori NJ. Articular cartilage friction increases in hip joints after the removal of acetabular labrum. J Biomech. 2012 Feb 2;45(3):524-30. doi: 10.1016/j.jbiomech.2011.11.044. Epub 2011 Dec 15. PMID 22176711
- [Background] Byrd JW. The role of hip arthroscopy in the athletic hip. Clin Sports Med. 2006 Apr;25(2):255-78, viii. doi: 10.1016/j.csm.2005.12.007. PMID 16638490
- [Background] Khanduja V, Villar RN. Arthroscopic surgery of the hip: current concepts and recent advances. J Bone Joint Surg Br. 2006 Dec;88(12):1557-66. doi: 10.1302/0301-620X.88B12.18584. PMID 17159164
- [Background] Kelly BT, Weiland DE, Schenker ML, Philippon MJ. Arthroscopic labral repair in the hip: surgical technique and review of the literature. Arthroscopy. 2005 Dec;21(12):1496-504. doi: 10.1016/j.arthro.2005.08.013. PMID 16376242
- [Background] Montgomery SR, Ngo SS, Hobson T, Nguyen S, Alluri R, Wang JC, Hame SL. Trends and demographics in hip arthroscopy in the United States. Arthroscopy. 2013 Apr;29(4):661-5. doi: 10.1016/j.arthro.2012.11.005. Epub 2013 Feb 1. PMID 23375668
- [Background] Fry R, Domb B. Labral base refixation in the hip: rationale and technique for an anatomic approach to labral repair. Arthroscopy. 2010 Sep;26(9 Suppl):S81-9. doi: 10.1016/j.arthro.2010.01.021. Epub 2010 Jul 7. PMID 20615651
- [Background] Lubowitz JH, Poehling GG. Watch your footprint: anatomic ACL reconstruction. Arthroscopy. 2009 Oct;25(10):1059-60. doi: 10.1016/j.arthro.2009.08.001. No abstract available. PMID 19801278
- [Background] Audenaert EA, Dhollander AA, Forsyth RG, Corten K, Verbruggen G, Pattyn C. Histologic assessment of acetabular labrum healing. Arthroscopy. 2012 Dec;28(12):1784-9. doi: 10.1016/j.arthro.2012.06.012. Epub 2012 Oct 17. PMID 23084152
- [Background] Philippon MJ, Arnoczky SP, Torrie A. Arthroscopic repair of the acetabular labrum: a histologic assessment of healing in an ovine model. Arthroscopy. 2007 Apr;23(4):376-80. doi: 10.1016/j.arthro.2007.01.017. PMID 17418329
- [Background] Petersen W, Petersen F, Tillmann B. Structure and vascularization of the acetabular labrum with regard to the pathogenesis and healing of labral lesions. Arch Orthop Trauma Surg. 2003 Jul;123(6):283-8. doi: 10.1007/s00402-003-0527-7. Epub 2003 Jun 7. PMID 12802599
- [Background] Syed HM, Martin SD. Arthroscopic acetabular recession with chondrolabral preservation. Am J Orthop (Belle Mead NJ). 2013 Apr;42(4):181-4. PMID 23630678
- [Background] Matles AL. A microscopic study of the newborn fibrocartilagenous acetabular labrum. Clin Orthop Relat Res. 1967 Sep-Oct;54:197-206. No abstract available. PMID 4173072
- [Background] Seldes RM, Tan V, Hunt J, Katz M, Winiarsky R, Fitzgerald RH Jr. Anatomy, histologic features, and vascularity of the adult acetabular labrum. Clin Orthop Relat Res. 2001 Jan;(382):232-40. doi: 10.1097/00003086-200101000-00031. PMID 11153993
- [Background] Lohe F, Eckstein F, Sauer T, Putz R. Structure, strain and function of the transverse acetabular ligament. Acta Anat (Basel). 1996;157(4):315-23. doi: 10.1159/000147894. PMID 9259881
- [Background] Konrath GA, Hamel AJ, Olson SA, Bay B, Sharkey NA. The role of the acetabular labrum and the transverse acetabular ligament in load transmission in the hip. J Bone Joint Surg Am. 1998 Dec;80(12):1781-8. doi: 10.2106/00004623-199812000-00008. PMID 9875936
- [Background] Cashin M, Uhthoff H, O'Neill M, Beaule PE. Embryology of the acetabular labral-chondral complex. J Bone Joint Surg Br. 2008 Aug;90(8):1019-24. doi: 10.1302/0301-620X.90B8.20161. PMID 18669956
- [Background] Bedi A, Kelly BT. Femoroacetabular impingement. J Bone Joint Surg Am. 2013 Jan 2;95(1):82-92. doi: 10.2106/JBJS.K.01219. PMID 23283377
- [Background] McCarthy JC. The diagnosis and treatment of labral and chondral injuries. Instr Course Lect. 2004;53:573-7. PMID 15116646
- [Background] Ferguson SJ, Bryant JT, Ganz R, Ito K. The influence of the acetabular labrum on hip joint cartilage consolidation: a poroelastic finite element model. J Biomech. 2000 Aug;33(8):953-60. doi: 10.1016/s0021-9290(00)00042-7. PMID 10828325
- [Background] Ferguson SJ, Bryant JT, Ganz R, Ito K. The acetabular labrum seal: a poroelastic finite element model. Clin Biomech (Bristol). 2000 Jul;15(6):463-8. doi: 10.1016/s0268-0033(99)00099-6. PMID 10771126
- [Background] Ferguson SJ, Bryant JT, Ganz R, Ito K. An in vitro investigation of the acetabular labral seal in hip joint mechanics. J Biomech. 2003 Feb;36(2):171-8. doi: 10.1016/s0021-9290(02)00365-2. PMID 12547354
- [Background] Larson CM, Giveans MR. Arthroscopic debridement versus refixation of the acetabular labrum associated with femoroacetabular impingement. Arthroscopy. 2009 Apr;25(4):369-76. doi: 10.1016/j.arthro.2008.12.014. Epub 2009 Mar 5. PMID 19341923
- [Background] Espinosa N, Beck M, Rothenfluh DA, Ganz R, Leunig M. Treatment of femoro-acetabular impingement: preliminary results of labral refixation. Surgical technique. J Bone Joint Surg Am. 2007 Mar;89 Suppl 2 Pt.1:36-53. doi: 10.2106/JBJS.F.01123. PMID 17332124
- [Background] Larson CM, Giveans MR, Stone RM. Arthroscopic debridement versus refixation of the acetabular labrum associated with femoroacetabular impingement: mean 3.5-year follow-up. Am J Sports Med. 2012 May;40(5):1015-21. doi: 10.1177/0363546511434578. Epub 2012 Feb 3. PMID 22307078
- [Background] Limbird TJ. Application of laser Doppler technology to meniscal injuries. Clin Orthop Relat Res. 1990 Mar;(252):88-91. PMID 2406079
- [Background] Perimed. Laser Doppler Probes. Perimed AB. Web. 25 Aug. 2013.
- [Background] Levy O, Relwani J, Zaman T, Even T, Venkateswaran B, Copeland S. Measurement of blood flow in the rotator cuff using laser Doppler flowmetry. J Bone Joint Surg Br. 2008 Jul;90(7):893-8. doi: 10.1302/0301-620X.90B7.19918. PMID 18591599
- [Background] Swiontkowski MF, Schlehr F, Sanders R, Limbird TA, Pou A, Collins JC. Direct, real time measurement of meniscal blood flow. An experimental investigation in sheep. Am J Sports Med. 1988 Sep-Oct;16(5):429-33. doi: 10.1177/036354658801600501. PMID 3189673
- [Background] Swiontkowski MF, Iannotti JP, Boulas HJ, Esterhai JL. Intraoperative assessment of rotator cuff vascularity using laser doppler flowmetry. In: Post M, Morr, eds. Surgery of the shoulder. St. Louis: Mosby, 1990: 208-12.
- [Background] Rathbun JB, Macnab I. The microvascular pattern of the rotator cuff. J Bone Joint Surg Br. 1970 Aug;52(3):540-53. No abstract available. PMID 5455089
- [Background] McCarthy JC, Jarrett BT, Ojeifo O, Lee JA, Bragdon CR. What factors influence long-term survivorship after hip arthroscopy? Clin Orthop Relat Res. 2011 Feb;469(2):362-71. doi: 10.1007/s11999-010-1559-2. PMID 20872105
- [Background] Hettrich CM, Crawford D, Rodeo SA. Cartilage repair: third-generation cell-based technologies--basic science, surgical techniques, clinical outcomes. Sports Med Arthrosc Rev. 2008 Dec;16(4):230-5. doi: 10.1097/JSA.0b013e31818cdc98. PMID 19011555
- [Background] Holton J, Imam MA, Snow M. Bone Marrow Aspirate in the Treatment of Chondral Injuries. Front Surg. 2016 Jun 16;3:33. doi: 10.3389/fsurg.2016.00033. eCollection 2016. PMID 27379241
- [Background] Green CJ, Beck A, Wood D, Zheng MH. The biology and clinical evidence of microfracture in hip preservation surgery. J Hip Preserv Surg. 2016 Feb 26;3(2):108-23. doi: 10.1093/jhps/hnw007. eCollection 2016 Jul. PMID 27583147
- [Background] Jordan MA, Van Thiel GS, Chahal J, Nho SJ. Operative treatment of chondral defects in the hip joint: a systematic review. Curr Rev Musculoskelet Med. 2012 Sep;5(3):244-53. doi: 10.1007/s12178-012-9134-y. PMID 22814674
- [Background] Dhollander AA, De Neve F, Almqvist KF, Verdonk R, Lambrecht S, Elewaut D, Verbruggen G, Verdonk PC. Autologous matrix-induced chondrogenesis combined with platelet-rich plasma gel: technical description and a five pilot patients report. Knee Surg Sports Traumatol Arthrosc. 2011 Apr;19(4):536-42. doi: 10.1007/s00167-010-1337-4. Epub 2010 Dec 11. PMID 21153540
- [Background] Murrell WD, Anz AW, Badsha H, Bennett WF, Boykin RE, Caplan AI. Regenerative treatments to enhance orthopedic surgical outcome. PM R. 2015 Apr;7(4 Suppl):S41-S52. doi: 10.1016/j.pmrj.2015.01.015. PMID 25864660
- [Background] Hernigou P, Flouzat Lachaniette CH, Delambre J, Zilber S, Duffiet P, Chevallier N, Rouard H. Biologic augmentation of rotator cuff repair with mesenchymal stem cells during arthroscopy improves healing and prevents further tears: a case-controlled study. Int Orthop. 2014 Sep;38(9):1811-8. doi: 10.1007/s00264-014-2391-1. Epub 2014 Jun 7. PMID 24913770
- [Background] Ellera Gomes JL, da Silva RC, Silla LM, Abreu MR, Pellanda R. Conventional rotator cuff repair complemented by the aid of mononuclear autologous stem cells. Knee Surg Sports Traumatol Arthrosc. 2012 Feb;20(2):373-7. doi: 10.1007/s00167-011-1607-9. Epub 2011 Jul 20. PMID 21773831
- [Background] Kanaya A, Deie M, Adachi N, Nishimori M, Yanada S, Ochi M. Intra-articular injection of mesenchymal stromal cells in partially torn anterior cruciate ligaments in a rat model. Arthroscopy. 2007 Jun;23(6):610-7. doi: 10.1016/j.arthro.2007.01.013. PMID 17560475
- [Background] Filardo G, Perdisa F, Roffi A, Marcacci M, Kon E. Stem cells in articular cartilage regeneration. J Orthop Surg Res. 2016 Apr 12;11:42. doi: 10.1186/s13018-016-0378-x. PMID 27072345
- [Background] Emara KM, Diab RA, Emara AK. Recent biological trends in management of fracture non-union. World J Orthop. 2015 Sep 18;6(8):623-8. doi: 10.5312/wjo.v6.i8.623. eCollection 2015 Sep 18. PMID 26396938
- [Background] Kemp JL, Collins NJ, Roos EM, Crossley KM. Psychometric properties of patient-reported outcome measures for hip arthroscopic surgery. Am J Sports Med. 2013 Sep;41(9):2065-73. doi: 10.1177/0363546513494173. Epub 2013 Jul 8. PMID 23835268